CLINICAL TRIAL: NCT00356629
Title: Development of a Noninvasive Method of Evaluation of the Pulmonary Inflammation in the Condensates of Exhaled Air
Brief Title: Development of a Noninvasive Method of Evaluation of Pulmonary Inflammation in the Condensates of Exhaled Air
Status: Terminated | Type: Observational
Why Stopped: Technical problem
Sponsor: University Hospital, Tours (Other)
Responsible Party: University Hospital Tours/Jocelyne Marlière, University Hospital Tours
Other Study IDs: AOHP06-PD Air Exhalé
Record Dates: First submitted 2006-07-25; First posted 2006-07-26 (Estimated); Last update posted 2008-11-14 (Estimated); Status verified 2008-11

CONDITIONS: Bronchopulmonary Ignition; Condensate of Exhaled Air; Mucoviscidosis; Asthma
Keywords: bronchopulmonary ignition; condensate of exhaled air; Mucoviscidosis; Asthma
MeSH Terms: conditions — Cystic Fibrosis; Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the study is identify biological parameters reflecting proteolytic activity in the exhaled condenstaes which might be useful to follow up pulmonary inflammation in various conditions including cystic fibrosis, COPD, asthma, tobacco exposure. Three proteases will be analyzed, i.e. elastase, proteinase 3 and cathepsin G. Results in the condensates will be compared to those obtained in sputum.

DETAILED DESCRIPTION:
5 groups of 20 individuals each: group 1 CF, group 2 COPD, group 3 asthma, group 4 tobacco exposure, group 5 control subjects.

Collection of exhaled condensates in all subjects and of sputum in subjects belonging to groups 1 and 2.

Clinical examination and PFTs in all patients.

ELIGIBILITY:
Inclusion criteria

* Subjects suffering from CF, COPD, asthma and tobacco exposure (groups 1 to 4) and controls (group 5)
* aged more or equal to 18
* stable disease
* able to perform PFTs
* informed consent signed
* affiliated to french social insurance

Exclusion Criteria:

* acute exacerbation of the disease during the last 2 weeks
* IV or oral steroids or antibiotics during the last 2 weeks
* hospitalization during the last 2 weeks
* colonization by S aureus methicillin resistant and/or Burkholderia cepacia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ubjects suffering from CF, COPD, asthma and tobacco exposure
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2006-07; Study Completion 2008-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: DIOT Patrice, Pr, Principal Investigator — service de Pneumologie et EFR CHRU Tours
Locations (1):
- Service de Pneumologie et EFR CHRU Tours, Tours, France

REFERENCES:
- [Background] Attucci S, Gauthier A, Korkmaz B, Delepine P, Martino MF, Saudubray F, Diot P, Gauthier F. EPI-hNE4, a proteolysis-resistant inhibitor of human neutrophil elastase and potential anti-inflammatory drug for treating cystic fibrosis. J Pharmacol Exp Ther. 2006 Aug;318(2):803-9. doi: 10.1124/jpet.106.103440. Epub 2006 Apr 20. PMID 16627747
- [Background] Grimbert D, Vecellio L, Delepine P, Attucci S, Boissinot E, Poncin A, Gauthier F, Valat C, Saudubray F, Antonioz P, Diot P. Characteristics of EPI-hNE4 aerosol: a new elastase inhibitor for treatment of cystic fibrosis. J Aerosol Med. 2003 Summer;16(2):121-9. doi: 10.1089/089426803321919889. PMID 12823906
- See also: Related Info — http://u618.univ-tours.fr